CLINICAL TRIAL: NCT07258875
Title: Effect of VExUS Ultrasound Protocol (Venous Excess Ultrasound) on Perioperative Fluid Management, on the Incidence of Postoperative Pulmonary Complications and Postoperative Acute Kidney Injury in Patients Undergoing Thoracic Surgery
Acronym: VEXUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Alexandros Bogas, Alexandros Bogas Manouselis, University of Crete
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18721
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Thoracic Surgery With One-lung Ventilation; VExUS; Fluid Management; Acute Kidney Injury; Postoperative Pulmonary Complications (PPCs)
Keywords: VExUS, fluid management, pulmonary complications, acute kidney injury, thoracic surgery, one lung ventilation
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A single-center clinical study conducted in the Anesthesiology Clinic of the University General Hospital of Heraklion.
  Parallel design in two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care group (Placebo Comparator): Intraoperatively patients of the control group will be administered isotonic crystalloids (Lactated Ringer's, Plasma-Lyte) at a rate of 3 mL/kg/h.Fluid administration will continue at a rate of 3 mL/kg/h as per standard practice in the postanaesthesia care unit( PACU) also.In both groups, blood losses more than 300 ml will be replaced with a 5% albumin solution at a 1:1 ratio. Transfusion will be administered to maintain hemoglobin levels at 9 mg/dL. Both groups will follow the same multimodal anesthesia-analgesia protocol, with restricted opioid use in accordance with the departmental routine.
  Intraoperative hypotension (systolic arterial pressure < 90 mmHg or a decrease > 20% from baseline) will be managed with titrated norepinephrine infusion.
  Interventions: Other: Standard of Care (SOC)
- vexus guided group (Active Comparator): The VExUS evaluation will be performed pre- and immediately post-intubation before one-lung ventilation initiation.
  Ultrasound monitoring will be performed according to the VExUS protocol before positioning the patient in the lateral decubitus position. In patients with VExUS grade 0, a bolus of 250-500 mL (approximately 3 mL/kg) will be administered, followed by the infusion of crystalloids at a rate of 3 mL/kg/h. The inferior vena cava (IVC) diameter will be measured three times: once prior to anesthesia induction, once immediately after intubation, and once before patient emergence from anesthesia. In patients with VExUS grade 1, no bolus will be given, and only a fluid infusion at 3 mL/kg/h will be administered. In patients with VExUS grades 2 and 3, 10 mg of furosemide will be administered intravenously, followed by crystalloids infusion at a rate of 2 mL/kg/h.VExUS ultrasound will be repeated postoperatively in the PACU, following the same pattern of intervention.
  Interventions: Diagnostic Test: Venous Excess Ultrasound

INTERVENTIONS:
Diagnostic Test: Venous Excess Ultrasound — The VExUS protocol is a standardized point-of-care ultrasound examination that includes measurements of the inferior vena cava (IVC) diameter, combined with Doppler analysis of waveforms in the hepatic vein, portal vein, and renal veins. From this analysis, the presence of venous congestion-classified as mild or severe-or its absence is determined. A high VExUS score (grade 3) has been strongly associated with the occurrence of acute kidney injury in patients undergoing cardiac surgery and has more recently been linked to elevated right atrial pressure (RAP ≥ 12 mmHg). The protocol includes the following classification:
  * Grade 0: IVC < 2 cm
  * Grade 1: IVC ≥ 2 cm, with normal or mildly abnormal waveforms in the hepatic, portal, and renal veins (mild congestion)
  * Grade 2: IVC ≥ 2 cm, with severely altered waveforms in at least one vein (moderate congestion)
  * Grade 3: IVC ≥ 2 cm, with severely altered waveforms in multiple veins (severe congestion)
  Other Names: VEXUS
  Arms: vexus guided group
Other: Standard of Care (SOC) — Intraoperatively patients of the control group will be administered isotonic crystalloids (Lactated Ringer's, Plasma-Lyte) at a rate of 3 mL/kg/h.Fluid administration will continue at a rate of 3 mL/kg/h as per standard practice in the PACU.
  Other Names: standard of care
  Arms: standard of care group

SUMMARY:
This study aims to investigate the effect of a VExUS ultrasound guided protocol of perioperative fluid management within a goal-directed therapy framework, on postoperative respiratory complications, and the occurrence of acute kidney injury (AKI) in patients undergoing thoracic surgery.

DETAILED DESCRIPTION:
In thoracic surgery, intraoperative fluid management presents a challenge for anesthesiologists, as patients are at high risk of developing interstitial and alveolar edema of the lungs. A history of pulmonary disease, previous chemotherapy or radiation therapy in the area, one-lung ventilation, surgical manipulation, and ischemia-reperfusion injury can all damage the respiratory epithelium's glycocalyx, the alveolar epithelium, and surfactant, ultimately leading to pulmonary injury. These factors, combined with liberal perioperative fluid management, increase the risk of acute respiratory distress syndrome (ARDS), atelectasis, pneumonia, and ultimately postoperative mortality. Traditionally, a restrictive fluid management strategy is employed intraoperatively, with crystalloid administration at a rate of 1-2 ml/kg/h, ensuring that the perioperative fluid balance does not exceed 1500 ml. This restrictive strategy may increase the risk of hypovolemia, which can lead to tissue hypoperfusion, target organ dysfunction, and acute kidney injury. Within the Enhanced Recovery After Surgery (ERAS) protocols, goal-directed therapy (GDT) for fluid management in thoracic surgery is discussed but not explicitly recommended. Recommendations include avoiding overly restrictive or completely liberal fluid strategies, maintaining euvolemia, and preventing tissue hypoperfusion with balanced use of inotropic agents and fluid administration.

Pulmonary injury is the leading cause of death following thoracic surgery. Pre-existing respiratory disease, surgical manipulation, lung parenchyma resection, and the detrimental effects of one-lung ventilation increase the risk of postoperative respiratory complications. Although overhydration and ventilation with high tidal volumes have been replaced by a restrictive fluid strategy and the application of protective mechanical ventilation, it appears that all factors involved in ventilator-induced lung injury (VILI) also play a harmful role in one-lung ventilation. High strain on the ventilated lung, oxidative stress, surgical trauma, recruitment maneuvers, biological trauma, atelectatic trauma, and ischemia-reperfusion injury are the pathophysiological mechanisms leading to postoperative acute respiratory failure and, in 2-5% of cases, to ARDS.

Postoperative acute kidney injury (AKI) represents 18-47% of in-hospital AKI and is associated with prolonged hospitalization and high morbidity and mortality. Recently, the implementation of new AKI classifications (RIFLE, AKIN, KDIGO) has facilitated its early recognition for immediate preventive measures. Additionally, the detection of two early urinary biomarkers of kidney stress, the tissue inhibitor of metalloproteinases-2 (TIMP-2) and the insulin-like growth factor-binding protein 7 (IGFBP7), has contributed to this. Postoperatively, an increase in serum creatinine by up to 0.5 mg/dL from baseline has been associated with a threefold increase in mortality following cardiac surgery. Potential pathophysiological mechanisms of postoperative AKI include ischemia, inflammation, and toxins. However, in thoracic surgeries, both the hypovolemia of a restrictive fluid administration strategy and overhydration and venous congestion can equally lead to acute kidney injury postoperatively.

The VExUS protocol is a standardized point-of-care ultrasound examination that includes measurements of the inferior vena cava (IVC) diameter, combined with Doppler analysis of waveforms in the hepatic vein, portal vein, and renal veins. From this analysis, the presence of venous congestion-classified as mild or severe-or its absence is determined. A high VExUS score (grade 3) has been strongly associated with the occurrence of acute kidney injury in patients undergoing cardiac surgery and has more recently been linked to elevated right atrial pressure (RAP ≥ 12 mmHg). The protocol includes the following classification:

Grade 0: IVC < 2 cm Grade 1: IVC ≥ 2 cm, with normal or mildly abnormal waveforms in the hepatic, portal, and renal veins (mild congestion) Grade 2: IVC ≥ 2 cm, with severely altered waveforms in at least one vein (moderate congestion) Grade 3: IVC ≥ 2 cm, with severely altered waveforms in multiple veins (severe congestion).

A single-center clinical study conducted in the Anesthesiology Clinic of the University General Hospital of Heraklion.

Parallel design in two groups.Preoperative assessment, fasting, and premedication according to the routine of the department:

* Discontinuation of fluid intake 2 hours before surgery
* cessation of food intake 6 hours preoperatively
* discontinuation on the day of surgery of ACE inhibitors, angiotensin receptor blockers, thiazide diuretics, and loop diuretics.

Upon entering the operating room, patients will be connected standard ASA monitors: 5 lead ECG, pulse oximetry (SpO2), non-invasive blood pressure measurement. Under local anaesthesia an arterial catheter will be placed for invasive blood pressure measurement and blood gas sampling, along with at least two venous catheters of 16-20 G. Anesthesia and postoperative analgesia management will depend solely on the discretion of the responsible anesthesiologist. After anesthesia induction and double-lumen endotracheal tube placement, patients will be connected to the anesthesia machine, recruitment maneuvers will be performed with PEEP titration, and they will be mechanically ventilated applying the principles of protective mechanical ventilation. The correct placement of the endotracheal tube will be confirmed with fiberoptic bronchoscopy immediately after placement. A urinary catheter will be placed for hourly urine measurement, along with a thermometer.

Intraoperatively, the total administered fluids, hourly urine output, type and dose of vasopressor medications, and blood pressure (SAP, DAP, MAP) will be recorded every 15 minutes (unless a significant change occurs), along with arterial blood gases and lactate.

Protective Mechanical Ventilation of One Lung:

Ventilated lung:

Tidal volume (Vt): 4-5 ml/kg ideal body weight, Appropriate PEEP of 5-15 cmH2O, possible repeat of recruitment maneuver Plateau pressure - PEEP: up to 15 cmH2O, Management of respiratory rate (RR) aiming for permitted mild hypercapnia (PaCO2 = 40-60 mmHg), Modification of the I ratio to avoid air trapping and the emergence of PEEPi, Titration of FiO2 to achieve SpO2 = 88-92%, Protection against hypoxic pulmonary vasoconstriction by avoiding vasodilators, hypoventilation, alkalosis, hypothermia, and if inhaled anesthetics are used, maintaining MAC < 1, Mechanical ventilation model: Volume Control- Auto Flow on the Perseus A500 and Atlan A350 machines from Drager available in the Anesthesia Clinic.

Non-ventilated lung with SpO2 < 88%:

Recruitment maneuvers with the use of PEEP if possible, Use of CPAP, FiO2 = 100% and cessation of one lung ventilation.

Control Group:

Intraoperatively patients of the control group will be administered isotonic crystalloids (Lactated Ringer's, Plasma-Lyte) at a rate of 3 mL/kg/h.

VExUS-guided Group:

VExUS Evaluation. The VExUS evaluation will be performed pre- and immediately post-intubation before one-lung ventilation initiation. A trained anesthesiologist (will evaluate the patient according to the VExUS protocol, measuring the IVC diameter and performing Doppler analysis of the hepatic, portal, and renal veins. A VExUS score will be assigned as outlined in the section above.

Ultrasound monitoring will be performed according to the VExUS protocol before positioning the patient in the lateral decubitus position. In patients with VExUS grade 0, a bolus of 250-500 mL (approximately 3 mL/kg) will be administered, followed by the infusion of crystalloids at a rate of 3 mL/kg/h. The inferior vena cava (IVC) diameter will be measured three times: once prior to anesthesia induction, once immediately after intubation, and once before patient emergence from anesthesia. In patients with VExUS grade 1, no bolus will be given, and only a fluid infusion at 3 mL/kg/h will be administered. In patients with VExUS grades 2 and 3, 10 mg of furosemide will be administered intravenously, followed by crystalloids infusion at a rate of 2 mL/kg/h.

In both groups, blood losses will be replaced with a 5% albumin solution at a 1:1 ratio. Transfusion will be administered to maintain hemoglobin levels at 9 mg/dL. Both groups will follow the same multimodal anesthesia-analgesia protocol, with restricted opioid use in accordance with the departmental routine.

Intraoperative hypotension (systolic arterial pressure < 90 mmHg or a decrease > 20% from baseline) will be managed with titrated norepinephrine infusion.

Post-Anesthesia Care Unit (PACU)

Control Group:

Fluid administration will continue at a rate of 3 mL/kg/h as per standard practice.

VExUS-guided Group:

VExUS ultrasound will be repeated postoperatively. In patients with VExUS grade 0, a bolus of 250-500 mL (approximately 3 mL/kg) will be administered, followed by the infusion of crystalloids at a rate of 3 mL/kg/h. In patients with grades 1 to 3, 10 mg of intravenous furosemide will be administered, followed by a fluid infusion at 3 mL/kg/h and reassessment.

Patients will be monitored daily for the occurrence of postoperative respiratory complications as defined by the European Society of Anaesthesiology. Preoperative blood gas values (PaO2, PaCO2) will be measured as baseline, and postoperative blood gases will be collected on the 1st and 3rd postoperative days in the PACU. Oxygenation will be assessed using the PaO2/FiO2 ratio, and lactate levels will be measured concurrently.

Additionally, for each patient, estimated glomerular filtration rate (eGFR) using serum creatinine, cystatin C or both will be calculated preoperatively and on the 1st and 3rd postoperative days in PACU. To assess acute kidney injury (AKI), serum creatinine and cystatin C will be measured on the 1st and 3rd postoperative days, and AKI diagnosis and classification will follow KDIGO (Kidney Disease Improving Global Outcomes) criteria.

The following kidney injury biomarkers will also be measured:

Serum cystatin C, Total urine protein and albumin, Urine beta-2 microglobulin, Urine creatinine. Kidney stress biomarkers TIMP-2 and IGFBP7 in urine, as described above, will be measured immediately postoperatively in the PACU.

These biomarkers will also be measured in the PACU and on the 1st and 3rd postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years undergoing video assisted thoracic surgery/ lobectomy requiring one-lung ventilation.

Exclusion Criteria:

* Refusal to participate.
* Pneumonectomy.
* Young athletes (risk of physiologically large IVC >2 cm).
* Moderate-severe tricuspid regurgitation, moderate to severe pulmonary hypertension
* Heart failure with reduced ejection fraction, EF<35%
* Portal hypertension, portal vein thrombosis, or liver cirrhosis.
* Stage 4 or end-stage chronic kidney disease (eGFR <30 mL/min/1.73 m² or dialysis).
* Transfusion with more than 2 packed red blood cells unit perioperatively (intraoperatively, in the PACU, in the ward)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Kidney function-estimated glomerular filtration rate preoperatively | preoperatively
  Estimated glomerular filtration rate (eGFR) using serum creatinine, cystatin C or both calculated by CKD-EPI 2021 and MDRD equation
Kidney function-estimated glomerular filtration rate in the PACU | in the PACU
  Estimated glomerular filtration rate (eGFR) using serum creatinine, cystatin C or both calculated by CKD-EPI 2021 and MDRD equation
Kidney function- estimated glomerular filtration rate on postoperative day 1 | postoperative day 1
  Estimated glomerular filtration rate (eGFR) using serum creatinine, cystatin C or both calculated by CKD-EPI 2021 or MDRD equation.
Kidney function-estimated glomerular filtration rate on postoperative day 3 | on postoperative day 3
  Estimated glomerular filtration rate (eGFR) using serum creatinine, cystatin C or both calculated by tha CKD-EPI 2021 and MDRD equation
Urine output intraoperatively | From anesthesia induction, until the end of surgery
  Kidney function as quantified by urine output. Data will be reported as an averaged intraoperative rate in ml/kg*h.
Urinary output postoperatively in the PACU | during the PACU stay
  Kidney function as quantified by urine output. Data will be reported as an averaged intraoperative rate in ml/kg*h.
Renal stress biomarkers TIMP-2,IGFBP-7 | postoperatively in the PACU
  The detection of two early urinary biomarkers of kidney stress, the tissue inhibitor of metalloproteinases-2 (TIMP-2) and the insulin-like growth factor-binding protein 7 (IGFBP7), has contributed to early diagnosis of AKI and renal stress.Urine sample collection will take place in both study groups.
Serum Creatinine preoperatively | preoperatively
  Baseline serum creatinine measurement, in mg/dl.Blood sample collection will take place in both study groups.
Serum creatinine in the PACU | during the PACU stay
  serum creatinine measurement, in mg/dl.Blood sample collection will take place in both study groups.
Serum creatinine on postoperative day 1 | postoperative day 1
  Serum creatine measurement in mg/dlBlood sample collection will take place in both study groups.
Serum creatinine on postoperative day 3 | postoperative day 3
  measurement of serum creatinine in mg/dl.Blood sample collection will take place in both study groups.
Serum cystatin C preoperatively | preoperatively
  baseline measurement of serum cystatin C in mg/L.Blood sample collection will take place in both study groups.
serum cyctatin C in the PACU | during the PACU stay
  measurement of serum cystatin C postopertively in the PACU.Blood sample collection will take place in both study groups.
serum cystatin C on postoperative day 1 | postoperative day 1
  measurement of serum cystatin C in mg/L.Blood sample collection will take place in both study groups.
serum cystatin C on postoperative day 3 | postoperative day 3
  measurement of serum cystatin C in mg/LBlood sample collection will take place in both study groups.
urine beta-2 microglobulin preoperatively | preoperatively
  baseline measurement of beta-2 microglobulin in urine, as a renal stress marker.Urine sample collection will take place in both study groups.
urine beta-2 microglobulin in the PACU | during the PACU stay
  measurement of beta-2 microglobuline in urine.Urine sample collection will take place in both study groups.
urine beta-2 microglobulin on postoperative day 1 | postoperative day 1
  measurement of beta-2 microglobulin in urine.Urine sample collection will take place in both study groups.
urine beta-2 microglobulin on postoperative day 3 | postoperative day 3
  measurement of beta-2 microglobulin in urine.Urine sample collection will take place in both study groups.
total urine protein preoperatively | preoperatively
  baseline total urine protein measurement in mg/L in both groups of patients
total urine protein in the PACU | during the PACU stay
  Measurement of total urine protein in mg/l in both groups of patients
total urine protein on postoperative day 1 | postoperative day 1
  total urine protein measurement in mg/L in both groups of patients
total urine protein on postoperative day 3 | postoperative day 3
  measurement of total urine protein in mg/L in both groups of patients
urine albumin preoperatively | preoperatively
  baseline measurement of urine albumin in both groups of patients
urine albumin in the PACU | during the PACU stay
  urine albumin measurement in both groups of patients
urine albumin on postoperative day 1 | postoperative day 1
  measurement of urine albumin in both groups of patients
urine albumin on postoperative day 3 | postoperative day 3
  measurement of urine albumin in both groups of patients
urine creatinine preoperatively | preoperatively
  urine creatinine baseline measurement in g/L in both groups of patients
urine creatinine in the PACU | during the PACU stay
  urine creatinine measurement in g/L in both groups of patients
urine creatinine on postoperative day 1 | postoperative day 1
  measurement of urine creatinine in g/l in both groups of patients
urine creatinine on postoperative day 3 | postoperative day 3
  measurement of urine creatinine in g/l in both groups of patients
urine albumin to creatinine ratio preoperatively | preoperatively
  baseline measurement of urine albumin to creatinine ratio in both groups of patients
urine albumin to creatinine ratio in the PACU | during the PACU stay
  measurement of urine albumin to creatinine ratio in both groups of patients
urine albumin to creatinine ratio on postoperative day 1 | postoperative day 1
  measurement of urine albumin to creatinine ratio in both groups of patients
urine albumin to creatinine ratio on postoperative day 3 | postoperative day 3
  measurement of urine albumin to creatinine ratio in both groups of patients
urine protein to creatinine ratio preoperatively | preoperatively
  baseline measurement of urine protein to creatinine ratio in both groups of patients
urine protein to creatinine ratio in the PACU | during the PACU stay
  measurement of protein to creatinine ratio in both groups of patients
urine protein to creatinine ratio on postoperative day 1 | postoperative day 1
  measurement of protein to creatinine ratio in both groups of patients
urine protein to creatinine ratio on postoperative day 3 | postoperative day 3
  measurement of protein to creatinine ratio in both groups of patients
pulse oximetry (SpO2) preoperatively | preoperatively
  baseline pulse oximetry measurement in both groups of patients
pulse oximetry (SpO2) intraoperatively | during one lung ventilation
  mean of pulse oximetry measurements in both groups of patients
pulse oximetry (SpO2) in the PACU | during the PACU stay
  mean of pulse oximetry measurements in both groups of patients
pulse oximetry (SpO2) on postoperative day 1 | postoperative day 1
  pulse oximetry measurement in both groups of patients
pulse oximetry (SpO2) on postoperative day 3 | postoperative day 3
  pulse oximetry measurement in both groups of patients
arterial oxygen saturation (SaO2) preoperatively | preoperatively
  baseline measurement of arterial oxygen saturation in both groups of patients by arterial blood gas analysis
arterial oxygen saturation (SaO2) intraoperatively | intraoperatively
  mean of measurement of arterial oxygen saturation in both groups of patients by arterial blood gas analysis
arterial oxygen saturation (SaO2) in the PACU | during the PACU stay
  mean of measurement of arterial oxygen saturation in both groups of patients by arterial blood gas analysis
arterial oxygen saturation (SaO2) on postoperative day 1 | postoperative day 1
  measurement of arterial oxygen saturation in both groups of patients by arterial blood gas analysis
arterial oxygen saturation (SaO2) on postoperative day 3 | postoperative day 3
  measurement of arterial oxygen saturation in both groups of patients by arterial blood gas analysis
arterial carbon dioxide partial pressure (PaCO2) preoperatively | preoperatively
  baseline measurement of arterial carbon dioxide partial pressure in mmHg in both groups of patients
arterial carbon dioxide partial pressure intraoperatively | intraoperatively
  mean of arterial carbon dioxide partial pressure measurements in mmHg in both groups of patients
arterial carbon dioxide partial pressure in the PACU | during the PACU stay
  mean of arterial carbon dioxide partial pressure measurements in mmHg in both groups of patients
arterial carbon dioxide partial pressure on postoperative day 1 | postoperative day 1
  arterial carbon dioxide partial pressure measurement in mmHg in both groups of patients
arterial carbon dioxide partial pressure on postoperative day 3 | postoperative day 3
  arterial carbon dioxide partial pressure measurement in mmHg in both groups of patients
arterial oxygen partial pressure (PaO2) preoperatively | preoperatively
  arterial oxygen partial pressure baseline measurement in mmHg in both groups of patients
arterial oxygen partial pressure (PaO2) intraoperatively | intraoperatively
  mean of arterial oxygen partial pressure measurements in mmHg in both groups of patients during one lung ventilation
arterial oxygen partial pressure (PaO2) in the PACU | during the PACU stay
  mean of arterial oxygen partial pressure measurements in mmHg in both groups of patients
arterial oxygen partial pressure (PaO2) on postoperative day 1 | postoperative day 1
  arterial oxygen partial pressure measurement in mmHg in both groups of patients
arterial oxygen partial pressure (PaO2) on postoperative day 3 | postoperative day 3
  arterial oxygen partial pressure measurement in mmHg in both groups of patients
arterial lactate measurement preoperatively | preoperatively
  baseline measurement of arterial lactate in mmol/L by arterial blood gas analysis in both groups of patients
arterial lactate measurement intraoperatively | intraoperatively
  mean of measurements of arterial lactate in mmol/L by arterial blood gas analysis in both groups of patients
arterial lactate measurement in the PACU | during the PACU stay
  mean of measurements of arterial lactate in mmol/L by arterial blood gas analysis in both groups of patients
arterial lactate measurement on postoperative day 1 | postoperative day 1
  measurement of arterial lactate in mmol/L by arterial blood gas analysis in both groups of patients
arterial lactate measurement on postoperative day 3 | postoperative day 3
  measurement of arterial lactate in mmol/L by arterial blood gas analysis in both groups of patients
oxygen partial pressure to fraction of oxygen in inspired air ratio (P/F ratio) in arterial blood preoperatively | preoperatively
  baseline measurement of P/F ratio by arterial blood gas analysis in both groups of patients
oxygen partial pressure to fraction of oxygen in inspired air ratio (P/F ratio) in arterial blood intraoperatively | intraoperatively
  mean of measurements of P/F ratio by arterial blood gas analysis in both groups of patients
oxygen partial pressure to fraction of oxygen in inspired air ratio (P/F ratio) in arterial blood in the PACU | during the PACU stay
  mean of measurements of P/F ratio by arterial blood gas analysis in both groups of patients
oxygen partial pressure to fraction of oxygen in inspired air ratio (P/F ratio) in arterial blood on postoperative day 1 | postoperative day 1
  measurement of P/F ratio by arterial blood gas analysis in both groups of patients
oxygen partial pressure to fraction of oxygen in inspired air ratio (P/F ratio) in arterial blood on postoperative day 3 | postoperative day 3
  measurement of P/F ratio by arterial blood gas analysis in both groups of patients
occurrence of postoperative pulmonary complications (PCCs) on postoperative day 1 | on postoperative day 1
  Patients will be monitored for the occurrence of postoperative respiratory complications as defined by the European Society of Anaesthesiology, including aspiration pneumonitis, respiratory failure, ARDS, pulmonary infection, atelectasis, cardiopulmonary edema, pleural infusion, pneumothorax, pulmonary infiltrates, prolonged air leakage, purulent pleuritis, pulmonary embolism, lung hemorrhage and bronchospasm.
  Chest radiography obtaining on postoperative day 1, arterial blood gas analysis as already mentioned and clinical findings such as respiratory rate, heart rate, blood pressure, temperature, airway secretions, Visual analog scale of dyspnea will help to identify the presence or not of PCCs.
occurrence of postoperative pulmonary complications (PCCs) on postoperative day 3 | on postoperative day 3
  Patients will be monitored for the occurrence of postoperative respiratory complications as defined by the European Society of Anaesthesiology, including aspiration pneumonitis, respiratory failure, ARDS, pulmonary infection, atelectasis, cardiopulmonary edema, pleural infusion, pneumothorax, pulmonary infiltrates, prolonged air leakage, purulent pleuritis, pulmonary embolism, lung hemorrhage and bronchospasm.
  Chest radiography obtaining on postoperative day 3 or earlier, arterial blood gas analysis as already mentioned and clinical findings such as respiratory rate, heart rate, blood pressure, temperature, airway secretions, Visual analog scale of dyspnea will help to identify the presence or not of PCCs.

SECONDARY OUTCOMES:
long term kidney impairment | from enrollment to day 30 approximately
  serum and urine creatinine, serum urea, urine albumin and protein and consequently albumin to creatinine ratio and protein to creatinine ratio will be measured approximately 30 days postoperative, to asses long term renal dysfunction after VATS lobectomy.
Noradrenaline equivalent dose | from the surgery onset to the discharge from the post anesthesia care unit
  Both groups maintained stable blood pressures with norepinephrine support as needed, but VExUS group showed more hemodynamic stability, concerning the measurements of cardiac output, cardiac index, stroke volume and stroke volume variation ( pulse contour analysis). As though, a larger noradrenaline amount as total dose and consequently, a bigger noradrenaline equivalent dose is expected to be given perioperatively in the control group of standard of care.
Length of stay - Hospital Discharge | From date of randomization (day before surgery) until the date of the discharge from the hospital
  Hospital length of stay will be reported in days.
intraoperative hypotension | Baseline: 5 minutes prior to anaesthesia induction. Intraoperative Hypotension: From anesthesia induction, until the end of surgery
  Intraoperative Hypotension (defined as MAP≤65mmHg or ≤80% of preoperative Baseline), with episodes lasting ≥1 minute. All patients will have a 5 minute preoperative MAP baseline, with measurements every 20 seconds. Intraoperative data will be compared to the mean preoperative 5 minute MPB baseline.
hemodynamic stability: pulse contour analysis monitoring | Baseline: 5 minutes prior to anaesthesia induction.From anesthesia induction, until the end of surgery
  During the operation, a cardiac output monitor with waveform analysis will be used, providing calculations every 20 seconds for CO, CI, SV, SVI, SVV, SAP, DAP, MAP, and PR, without any decisions regarding fluid administration being made based on these measurements. In the control group, fluid administration will be fixed at 3 ml/kg/h, while in the VExUS group, fluid administration will be guided by the ultrasound protocol. Episodes of hypotension will be managed accordingly with the administration of vasoconstrictive drugs.These data will be used to compare the hemodynamic stability between the two groups.
RBCs tranfusion, FFP transfusion, PLT tranfusion intraoperatively | From anesthesia induction, until the end of surgery
  Concentrated RBC, FFP, PLT unit requirements. Data will be reported in ml.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, Professor of Anaesthesiology, Study Chair — Medical School, University of Crete
Locations (1):
- University General Hospital of Heraklion, Heraklion, Crete, Greece

REFERENCES:
- [Result] Dharnidharka VR, Kwon C, Stevens G. Serum cystatin C is superior to serum creatinine as a marker of kidney function: a meta-analysis. Am J Kidney Dis. 2002 Aug;40(2):221-6. doi: 10.1053/ajkd.2002.34487. PMID 12148093
- [Result] 13. Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work vexusGroup. KDIGO Clinical Practice Guideline for Acute Kidney Injury. Kidney inter., Suppl. 2012; 2: 1-138.
- [Result] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Result] Longino A, Martin K, Leyba K, Siegel G, Gill E, Douglas IS, Burke J. Correlation between the VExUS score and right atrial pressure: a pilot prospective observational study. Crit Care. 2023 May 26;27(1):205. doi: 10.1186/s13054-023-04471-0. PMID 37237315
- [Result] Magin JC, Wrobel JR, An X, Acton J, Doyal A, Jia S, Krakowski JC, Schoenherr J, Serrano R, Flynn D, McLean D, Grant SA. Venous Excess Ultrasound (VExUS Grading to Assess Perioperative Fluid Status for Noncardiac Surgeries: a Prospective Observational Pilot Study. POCUS J. 2023 Nov 27;8(2):223-229. doi: 10.24908/pocus.v8i2.16792. eCollection 2023. PMID 38099161
- [Result] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297
- [Result] Romagnoli S, Ricci Z. Postoperative acute kidney injury. Minerva Anestesiol. 2015 Jun;81(6):684-96. Epub 2014 Jul 24. PMID 25057935
- [Result] Park M, Yoon S, Nam JS, Ahn HJ, Kim H, Kim HJ, Choi H, Kim HK, Blank RS, Yun SC, Lee DK, Yang M, Kim JA, Song I, Kim BR, Bahk JH, Kim J, Lee S, Choi IC, Oh YJ, Hwang W, Lim BG, Heo BY. Driving pressure-guided ventilation and postoperative pulmonary complications in thoracic surgery: a multicentre randomised clinical trial. Br J Anaesth. 2023 Jan;130(1):e106-e118. doi: 10.1016/j.bja.2022.06.037. Epub 2022 Aug 20. PMID 35995638
- [Result] Lohser J, Slinger P. Lung Injury After One-Lung Ventilation: A Review of the Pathophysiologic Mechanisms Affecting the Ventilated and the Collapsed Lung. Anesth Analg. 2015 Aug;121(2):302-18. doi: 10.1213/ANE.0000000000000808. PMID 26197368
- [Result] Arslantas MK, Kara HV, Tuncer BB, Yildizeli B, Yuksel M, Bostanci K, Bekiroglu N, Kararmaz A, Cinel I, Batirel HF. Effect of the amount of intraoperative fluid administration on postoperative pulmonary complications following anatomic lung resections. J Thorac Cardiovasc Surg. 2015 Jan;149(1):314-20, 321.e1. doi: 10.1016/j.jtcvs.2014.08.071. Epub 2014 Sep 18. PMID 25304302
- [Result] Tarbell JM. Shear stress and the endothelial transport barrier. Cardiovasc Res. 2010 Jul 15;87(2):320-30. doi: 10.1093/cvr/cvq146. Epub 2010 Jun 12. PMID 20543206
- [Result] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT07258875/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT07258875/ICF_001.pdf